CLINICAL TRIAL: NCT04251975
Title: Effect of Intervention With Continuous Positive Pressure (CPAP) on Nocturnal Blood Pressure (BP) in Patients With Masked Hypertension and Sleep Apnea
Brief Title: Masked Hypertensive Patients With Obstructive Sleep Apnea
Acronym: Masked-OSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: Principal Investigator, Ferran Barbe, Head of Pulmonology, Sociedad Española de Neumología y Cirugía Torácica
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2131-Masked-OSA
Record Dates: First submitted 2020-01-07; First posted 2020-02-05 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Obstructive Sleep Apnea; Masked Hypertension
Keywords: Obstructive sleep apnea; Masked hypertension
MeSH Terms: conditions — Sleep Apnea, Obstructive; Masked Hypertension | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: This is an open-label, parallel, prospective, randomized and controlled trial.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPAP treatment (Experimental): Group of patients who will receive CPAP treatment
  Interventions: Device: CPAP treatment
- Conservative measures (No Intervention): Group of patients who will receive conservative treatment based on hygienic-dietetic measures

INTERVENTIONS:
Device: CPAP treatment — In this group of patients (CPAP group) will be prescribed CPAP treatment at an optimal pressure. It will be performed a CPAP titration with an automatic or manual CPAP according to usual clinical practice
  Arms: CPAP treatment

SUMMARY:
The general objective is to evaluate the effect of continuous positive airway pressure (CPAP) treatment in patients with masked hypertension.

The secondary objectives are: i) To evaluate the prevalence of different circadian patterns of BP in ambulatory blood pressure monitoring (ABPM) (dipper / non-dipper); ii) To assess in these patients the relationship between compliance with CPAP treatment and the response to nocturnal BP; iii) To identify variables of the ABPM, and biomarkers that are related to the unfavourable pattern of nocturnal BP response in these patients treated with CPAP; iv) To evaluate the change in the profile of biomarkers with the treatment.

Methodology: Open, parallel, prospective, randomized and controlled study in which an ABPM will be performed in individuals with masked hypertension referred to the sleep unit and diagnosed of OSA (AHI≥ 30) without sleepiness (Epworth≤18).

A total of 64 subjects with OSA and masked hypertension will be recruited. It will be collected blood for the determination of biomarkers. Subsequently, they will be randomized to receive treatment with CPAP (32) or conservative treatment (32). After 3 months of initiation, ABPM and biological determinations will be repeated.

DETAILED DESCRIPTION:
Recruitment: It will be recruited subjects with masked hypertension. For that, normotensive subjects (Blood pressure (BP)<140/90mmHg in the office) referred to the sleep unit of the Hospital Santa Maria (Spain) who are diagnosed of severe OSA (AHI≥30) by a sleep study and who do not present significant somnolence (Epworth≤18) will be proposed to participate in the study. Then, it will be performed an ABPM during-24 hours, and those subjects with an abnormal ABPM results and normal BP in the office will be included, are those subjects called masked hypertensive.

Definition of the groups: Patients will be randomized to receive one of the following treatments:

1. CPAP: Patients who will receive CPAP treatment. The CPAP titration will be carried out with an automatic or manual CPAP according to usual clinical practice.
2. Conservative treatment: Patients who will receive conservative treatment based on hygienic-dietetic measures.

Randomization: It will be carried out with an automated platform

Duration of the treatment: All patients randomized to CPAP will begin treatment as soon as possible after randomization, and will continue treatment until the study ends (3 months).

Patients who interrupt treatment will be excluded from the study. ABPM and blood sample collection will be performed on all included patients at the beginning of the study and at 3 months under treatment (CPAP or conservative care).

Follow-up: All patients will be evaluated at the beginning of the study, at first month and at three months during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women over 18 years of age
2. Referred to the sleep unit for suspected OSA
3. Being masked hypertensive and presenting an AHI≥ 30 in the sleep study
4. Signature of the informed consent.

Exclusion Criteria:

1. Previous CPAP treatment
2. Significant somnolence defined by an Epworth Sleepiness Scale (ESS) score higher than 18
3. Psychophysical inability to complete questionnaires
4. Previous diagnosis or suspicion of another sleep disorder
5. Presence of more than 50% of central apneas or Cheyne-Stokes respiration
6. Having a serious chronic disease: neoplasia, renal failure, severe chronic obstructive pulmonary disease, chronic depression and other chronic limiting diseases
7. Medical history that may interfere with the objectives of the study or, in the opinion of the researcher, may compromise the conclusions
8. Any medical, social or geographical factor that may endanger the patient's compliance
9. Having a profession of high risk (professional driver).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Effect of CPAP treatment on BP in masked hypertensive patients with severe OSA | 3 years
  Change in mmHg in the blood pressure of the ambulatory blood pressure monitoring parameters after the treatment

SECONDARY OUTCOMES:
Prevalence of the different circadian BP patterns (dipper/no-dipper) in the ABPM of masked hypertensive subjects diagnosed with severe OSA without significant somnolence (Epworth≤18) | 3 years
  The prevalence of each circadian patterns will be calculated from the baseline ambulatory blood pressure monitoring data
Association between CPAP use and blood pressure change in ABPM | 3 years
  The relation between CPAP compliance (hours/night) and changes in mean nighttime BP (mmHg) between baseline and at 3-months in ABPM measurements will be assesed
Ambulatory blood pressure parameters that could be related to the response to CPAP treatment | 3 years
  Using all the ABPM variables we will proceed to the identification of variables that are related to the change in mean nocturnal BP in patients treated with CPAP
Changes in the biomarkers' profile (mRNAs) after CPAP treatment | 3 years
  Using the blood samples obtained in the baseline and 3 months visit it will be evaluated possible changes in the biomarkers profile after CPAP treatment.
  Learning Phase: complete profile analysis (754 miRNAs) will be carried out in 24 patients Learning Phase: complete profile analysis (754 miRNAs) will be carried out in 24 patients representative of the change in BP in treated patients. The miRNAs associated with the change in BP will be identified from the 754 miRNAs potentially present in serum and plasma.
  Validation Phase: Specific primers will be designed for the real-time PCR amplification of the genes for which we have found a significant association The miRNAs found will be analyzed after 3 months of treatment. Analysis of biomarkers. Immunoassay techniques will evaluate the following markers before and after treatment: angiotensin I, II and III, plasma renin activity, atrial natriuretic peptide (ANP), brain natriuretic peptide (BNP) and endogenous ouabain.

CONTACTS AND LOCATIONS:
Overall Officials: Ferran Barbé Illa, MD, Principal Investigator — CIBERES, SEPAR
Locations (1):
- Hospital Universitari Arnau de Vilanova, Lleida, Spain